CLINICAL TRIAL: NCT02082041
Title: Measurement of Blood Perfusion in Response to Loading in Patients With Wounds
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Tamara Reid Bush, Principal Investigator, Michigan State University
Other Study IDs: WOUND-MSU
Record Dates: First submitted 2014-03-04; First posted 2014-03-10 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Wound Formation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Wounds on leg

SUMMARY:
The purpose of this study is to monitor the skin blood flow in the lower leg, with different levels and types of applied loads. These loads will not be placed over the patient's wound nor will they be higher than loads the skin normally experiences in daily activities. The results of this research will help investigators understand the development of pressure ulcers, commonly known as bedsores and stasis ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if he/she has a wound on one or both legs.

Exclusion Criteria:

* under the age of 18
* individuals with mental illness
* individuals who are unable to sit for an hour
* individuals whose wound care method prohibits testing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with wounds on their legs, wound clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in perfusion | Cross-sectional, evaluation time frame is approximately 2 hours occuring at the time of enrollment
  Skin perfusion will be measured as different loads are applied to the leg.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Bush, PhD, Principal Investigator — Michigan State University
Locations (1):
- Sparrow Wound Clinic, Lansing, Michigan, United States